CLINICAL TRIAL: NCT03982121
Title: ISILI (In Situ Immunotherapy of LIver Metastases): An Openlabel, Dose-finding, Phase I Study of Intratumoral Ipilimumab and TLR4 Agonist GLA-SE in Combination With Systemic Nivolumab and Chemotherapy (FOLFOX Regimen) in Patients With Colorectal Liver Metastases.
Brief Title: Study of Intratumoral Ipilimumab and TLR4 Agonist GLA-SE in Combination With Systemic Nivolumab and Chemotherapy
Acronym: ISILI
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study never began because of withdrawal of the industrial partner
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-005020-14; 2017/2630 (Other: CSET number)
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Folfox protocol; Nivolumab; Ipilimumab; glucopyranosyl lipid-A

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label, dose-escalation combination phase 1 study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- A (Experimental): FOLFOX IV + NIVOLUMAB IV
  Interventions: Drug: FOLFOX regimen; Drug: Nivolumab
- B (Experimental): FOLFOX IV + GLA IT
  Interventions: Drug: FOLFOX regimen; Drug: GLA-SE
- C (Experimental): FOLFOX IV + IPILIMUMAB IT
  Interventions: Drug: FOLFOX regimen; Drug: Ipilimumab
- D (Experimental): FOLFOX IV + NIVOLUMAB IV + GLA IT
  Interventions: Drug: FOLFOX regimen; Drug: Nivolumab; Drug: GLA-SE
- E (Experimental): FOLFOX IV + NIVOLUMAB IV + IPILIMUMAB IT
  Interventions: Drug: FOLFOX regimen; Drug: Nivolumab; Drug: Ipilimumab
- F (Experimental): LFOX IV + NIVOLUMAB IV + GLA IT + IPILIMUMAB IT
  Interventions: Drug: FOLFOX regimen; Drug: Nivolumab; Drug: Ipilimumab; Drug: GLA-SE

INTERVENTIONS:
Drug: FOLFOX regimen — Oxaliplatin 85 mg/m² Leucovorin (LV) levogyre form (LLV) 200 mg/m² or dextro-levogyre (DL-LV) racemic mixture 400 mg/m²) Fluorouracil 2400 mg/m²
Drug: Nivolumab — Nivolumab 240 mg
  Arms: A; D; E; F
Drug: Ipilimumab — Ipilimumab 5 or 10 or 25 mg
  Arms: C; E; F
Drug: GLA-SE — GLA-SE 1 or 2 or 5 or 10 or 20 μg
  Arms: B; D; F

SUMMARY:
To determine the maximum tolerated dose (MTD), the recommended phase 2 dose (RP2D) and the toxicity profile (NCI CTCAE v5.0 and immune related adverse events) of i.t. administration of anti-CTLA4 antibody (ipilimumab) and TLR4 agonist (synthetic glucopyranosyl lipid A formulated in a stable emulsion [GLA-SE]) in colorectal LM (CRLM) in combination with intravenous (i.v.) administration of anti-PD-1 antibody (nivolumab) and chemotherapy (FOLFOX regimen).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal adenocarcinoma.
2. At least one CRLM

   * measurable according to RECIST 1.1,
   * at least >2 cm in maximal diameter,
   * visible on non-contrast enhanced computerized tomography (CT) scan or ultrasonography,
   * amenable to biopsy,
   * and amenable to percutaneous i.t. injection.
3. At least one other metastasis (controlateral CRLM or a distant visceral or lymph node metastasis)

   * measurable according to RECIST 1.1,
   * and amenable to biopsy.
4. Tumor lesions located in previously irradiated areas are considered measurable if disease progression has been demonstrated in such lesions.
5. Tumor liver involvement <50% on baseline CT scan.
6. Previous failure of active drug classes in mCRC (fluoropyrimidines, oxaliplatin, irinotecan, EGFR inhibitors [if wild-type RAS mCRC] and antiangiogenics).
7. Representative tumor specimens at the initial diagnosis of CRC (paraffin blocks (preferred) or at least 10 unstained slides), with the corresponding pathology report, if available.
8. Age >/=18 years.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
10. Expected life expectancy >3 months (no rapidly progressive disease).
11. Adequate organ functions:

    * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L (blood cell transfusions are allowed), absolute neutrophil count (ANC) ≥1.5 x 109/L, platelets ≥100 x 109/L
    * Serum creatinine ≤1.5 X upper limit of normal (ULN) or creatinine clearance (measured, or calculated per institutional standard) ≥50 mL/min for subject with creatinine levels >1.5 x institutional ULN (glomerular filtration rate can also be used in place of creatinine or creatinine clearance)
    * Serum total bilirubin ≤1.5 ULN or direct (unconjugated) bilirubin ≤ULN for subjects with total bilirubin levels >1.5 ULN
    * AST (SGOT) and ALT (SGPT) ≤5 ULN
    * Albumin >33 g/L
    * International normalized ratio (INR) or prothrombin time (PT) ≤1.5 ULN unless subject is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants
12. Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 24 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. Female subjects of childbearing potential should be willing to use two validated methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 7 months after the last dose of study medication (Reference Section 5.9.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
14. Sexually active male subjects unless surgically sterile, must agree to use condoms as an effective barrier method of contraception or abstain from heterosexual activity for the course of the study through 7 months after the last dose of study medication. It is recommended that their sexual partners use an effective contraceptive during the same period.
15. Signed informed consent.
16. Affiliation to or beneficiary of a social security system.

Exclusion Criteria:

1. Allergy or contraindication to oxaliplatin (including peripheral neuropathy [≥ grade 2]), fluorouracil (including known dihydropyrimidine dehydrogenase (DPD) deficiency) or leucovorin or to any other study drug.
2. Prior history of intolerance to full-dose FOLFOX regimen.
3. History of anterior organ transplantation, including allograft stem cell transplantation
4. History of interstitial lung disease
5. Patients eligible for curative-intent local therapies (e.g., surgery or thermablation).
6. Contraindication to percutaneous injection/biopsy (e.g., coagulation disorder, anticoagulant or antiaggregant therapy). Patients treated with low molecular weight heparin (LMWH) are eligible if they can interrupt their treatment for biopsies and i.t. injections.
7. Concomitant administration of any other anticancer therapy during the trial treatment period.
8. Prior chemotherapy, targeted therapy or radiation therapy within 2 weeks prior to study Day 1 or adverse events due to a previously administered agent that have not recovered (i.e., ≤ Grade 1) at baseline.
9. Immunodeficiency or systemic steroid therapy equivalent to prednisolone >10mg/day or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
10. Other malignancy within 2 years prior to enrollment with the exception of curatively treated basal-cell carcinoma of the skin, squamous-cell carcinoma of the skin, and/or curatively resected in situ cervical and/or in situ breast cancers.
11. Symptomatic active central nervous system metastases and/or carcinomatous meningitis.
12. Active automimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or asymptomatic asthma/atopy under topical/aerosol therapies would be an exception to this rule. Subjects who require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with stable hypothyroidism on hormone replacement or Sjogren's syndrome will not be excluded from the study. Patients with controlled type 1diabetes mellitus on a stable insulin regimen may be eligible for this study.
13. Active infection requiring systemic therapy.
14. Pregnancy or breastfeeding, or inadequate contraceptive method, or expectation to conceive children within the projected duration of the trial, starting with the pre-screening or screening visit through 7 months after the last dose of trial treatment.
15. Prior immunotherapy, including anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibodies (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
16. Clinically significant liver disease (i.e., with clinical, biological or morphological signs or symptoms of liver dysfunction, such as jaundice, hepatic encephalopathy, non-malignant ascites, radiological/endoscopic evidence of portal hypertension, biological evidence of liver insufficiency, etc.), including active viral, alcoholic, or other hepatitis, cirrhosis, severe oxaliplatin-induced sinusoidal obstruction syndrome (SOS) and inherited liver disease.
17. Known active Hepatitis B virus infection (e.g., HBsAg reactive) or Hepatitis C virus infection (e.g., HCV RNA [qualitative] is detected) and positive Hepatitis test results.
18. Known history of Human Immunodeficiency Virus (HIV) (HIV 1 and 2 antibodies) and positive HIV test results.
19. Administration of a live vaccine within 30 days prior to the first dose of trial treatment.
20. Any physical, psychological or social condition/reason that would preclude adequate follow-up or hamper patient's safety according to the investigator's opinion.
21. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | For all the cohorts, the DLT period to determine the MTD will be 28 days
  MTD will be determined based on the DLT definitions and identified as the maximum dose level at which less than 33% of DLT are observed in the evaluable patients.
Recommanded phase 2 dose (RP2D) | RP2D will be assessed on 8 weeks
  RP2D will be determined based on the MTD identified, on analysis of DLT defining events

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided